CLINICAL TRIAL: NCT00549783
Title: BOTOX® Economic Spasticity Trial (BEST)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AGN/HO/SPA/001-191622
Record Dates: First submitted 2007-10-24; First posted 2007-10-26 (Estimated); Results first posted 2012-08-22 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-07

CONDITIONS: Muscle Spasticity
MeSH Terms: conditions — Muscle Spasticity | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum toxin type A 900kD (Active Comparator): First intra-muscular injection at the Baseline visit, and optional second injection of the randomised treatment after a minimum of 12 weeks to a maximum of 24 weeks following the Baseline visit.
  Interventions: Biological: Botulinum Toxin Type A 900kD
- Placebo (Placebo Comparator): First intra-muscular injection at the Baseline visit, and optional second injection of the randomised treatment after a minimum of 12 weeks to a maximum of 24 weeks following the Baseline visit.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Botulinum Toxin Type A 900kD — The exact dosage and number of injection sites is based on the size, number, and location of muscles involved; the severity of spasticity; and the presence of local muscle weakness.
  First intra-muscular injection at the Baseline visit, and optional second injection of the randomised treatment after a minimum of 12 weeks to a maximum of 24 weeks following the Baseline visit.
  Other Names: BOTOX®
  Arms: Botulinum toxin type A 900kD
Biological: Placebo — The exact dosage and number of injection sites is based on the size, number, and location of muscles involved; the severity of spasticity; and the presence of local muscle weakness.
  First intra-muscular injection at the Baseline visit, and optional second injection of the randomised treatment after a minimum of 12 weeks to a maximum of 24 weeks following the Baseline visit.
  Arms: Placebo

SUMMARY:
This is a study to investigate if patients who have had a stroke and suffer from spasticity might benefit from being given BOTOX® in addition to the normal Standard Care. Spasticity is characterized by stiffness or frequent cramps accompanied by pain and abnormal movements and can prevent the carrying out of everyday tasks such as walking and getting dressed. BOTOX® is a neurotoxin, which is used to prevent the contraction of muscle fibre and has been shown to reduce spasticity significantly. Patients will be enrolled in this study at about 33 locations in Europe and Canada. Study participation will last for about 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stroke due to a primary cerebral hemorrhage/infarction
* Subarachnoid hemorrhage producing an upper motor syndrome affecting one body side which results in a hemi-paralysis/plegia

Exclusion Criteria:

* Patients with fixed contracture as a result of spasticity in the upper or lower limb planned to be treated and/or patients with other causes of spasticity (e.g. multiple sclerosis, spinal cord injury, etc.)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2007-10; Primary Completion 2010-01 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (4):
- Edmonton, Alberta, Canada
- Beelitz, Germany
- Uppsala, Sweden
- Burslem, Stoke-on-Trent, United Kingdom

REFERENCES:
- [Derived] Borg J, Ward AB, Wissel J, Kulkarni J, Sakel M, Ertzgaard P, Akerlund P, Reuter I, Herrmann C, Satkunam L, Wein T, Girod I, Wright N; BEST Study Group. Rationale and design of a multicentre, double-blind, prospective, randomized, European and Canadian study: evaluating patient outcomes and costs of managing adults with post-stroke focal spasticity. J Rehabil Med. 2011 Jan;43(1):15-22. doi: 10.2340/16501977-0663. PMID 21174051

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Botulinum Toxin Type A 900kD | Placebo
Started | 139 | 135
Completed | 131 | 122
Not Completed | 8 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin Type A 900kD | Placebo | Total
Number analyzed (Participants) | 139 | 135 | 274
Age Continuous [Median (Full Range); unit: years] | 64.11 [22.6 to 81.2] | 61.86 [26.8 to 82.4] | 62.60 [22.6 to 82.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 59 | 113
  Male | 85 | 76 | 161

OUTCOME MEASURES:

1. Primary Outcome: Physician Assessment of Success, as Determined by Percentage of Patients Who Achieve Their Principal Active Functional Goal at Week 24
Description: Physician assessment of success, as determined by percentage of patients who achieve their principal active functional goal (i.e. a score of 0 to +2 inclusive on the goal attainment scale [GAS]) at week 24 (or 10 weeks post second injection). The GAS is a 6-point scale where -3 means function is worse than at start, 0 means the expected goal was attained, and +2 is much better function than expected.
Time Frame: Week 24
Population: Intent-to-treat, which consists of all patients who were randomized (started study) and received a baseline injection.
Measure: Number; unit: Percentage of Patients
Arm/Group | Botulinum Toxin Type A 900kD | Placebo
Number analyzed (Participants) | 139 | 134
Percentage of Patients | 40.9 | 33.3

2. Secondary Outcome: Physician Assessment of Success, as Determined by Percentage of Patients Who Achieve Their Principal Functional Goal at Week 12
Description: Physician assessment of success, as determined by percentage of patients who achieve their principal functional goal (i.e., a score of 0 to +2 inclusive on the goal attainment scale [GAS]) at week 12. The GAS is 6-point scale where -3 means function is worse than at start, 0 means the expected goal was attained, and +2 is much better function than expected.
Time Frame: Week 12
Population: Intent-to-treat, which consists of all patients who were randomized (started study) and received a baseline injection.
Measure: Number; unit: Percentage of Patients
Arm/Group | Botulinum Toxin Type A 900kD | Placebo
Number analyzed (Participants) | 139 | 134
Percentage of Patients | 33.1 | 28.9

3. Secondary Outcome: Physician Assessment of Success, as Determined by Percentage of Patients Who Achieve Their Principal Functional Goal at Week 52
Description: Physician assessment of success, as determined by percentage of patients who achieve their principal functional goal (i.e., a score of 0 to +2 inclusive on the goal attainment scale [GAS]) at week 52. The GAS is a 6-point scale where -3 means function is worse than at start, 0 means the expected goal was attained, and +2 is much better function than expected
Time Frame: Week 52
Population: Intent-to-treat, which consists of all patients who were randomized (started study) and received a baseline injection.
Measure: Number; unit: Percentage of Patients
Arm/Group | Botulinum Toxin Type A 900kD | Placebo
Number analyzed (Participants) | 139 | 134
Percentage of Patients | 45.0 | 52.4

4. Secondary Outcome: Patient Assessment of Success, as Determined by Percentage of Patients Who Achieve Their Principal Functional Goal at Week 12
Description: Patient assessment of success, as determined by percentage of patients who achieve their principal functional goal (i.e., a score of 0 to +2 inclusive on the goal attainment scale [GAS]) at week 12. The GAS is a 6-point scale where -3 means function is worse than at start, 0 means the expected goal was attained, and +2 is much better function than expected.
Time Frame: Week 12
Population: Intent-to-treat, which consists of all patients who were randomized (started study) and received a baseline injection.
Measure: Number; unit: Percentage of Patients
Arm/Group | Botulinum Toxin Type A 900kD | Placebo
Number analyzed (Participants) | 139 | 134
Percentage of Patients | 33.1 | 27.3

5. Secondary Outcome: Patient Assessment of Success, as Determined by Percentage of Patients Who Achieve Their Principal Functional Goal at Week 24
Description: Patient assessment of success, as determined by percentage of patients who achieve their principal functional goal (i.e., a score of 0 to +2 inclusive on the goal attainment scale [GAS]) at week 24 (or 10 weeks post second injection). The GAS is a 6-point scale where -3 means function is worse than at start, 0 means the expected goal was attained, and +2 is much better function than expected.
Time Frame: Week 24
Population: Intent-to-treat, which consists of all patients who were randomized (started study) and received a baseline injection.
Measure: Number; unit: Percentage of Patients
Arm/Group | Botulinum Toxin Type A 900kD | Placebo
Number analyzed (Participants) | 139 | 134
Percentage of Patients | 40.7 | 39.0

6. Secondary Outcome: Patient Assessment of Success, as Determined by Percentage of Patients Who Achieve Their Principal Functional Goal at Week 52
Description: Patient assessment of success, as determined by percentage of patients who achieve their principal functional goal (i.e., a score of 0 to +2 inclusive on the goal attainment scale [GAS]) at week 52. The GAS is a 6-point scale where -3 means function is worse than at start, 0 means the expected goal was attained, and +2 is much better function than expected.
Time Frame: Week 52
Population: Intent-to-treat, which consists of all patients who were randomized (started study) and received a baseline injection.
Measure: Number; unit: Percentage of Patients
Arm/Group | Botulinum Toxin Type A 900kD | Placebo
Number analyzed (Participants) | 139 | 134
Percentage of Patients | 48.9 | 50.8

7. Secondary Outcome: Activities of Daily Living Quality of Life (QOL) Score at Week 12
Description: Activities of Daily Living QOL score at week 12 as measured by SF-12 Physical Component (PCS-12). The SF-12 consists of 12 questions on various health questions. The PCS-12 is a sub-score calculated from the SF-12 total score based on the physical health questions where 0 is worse and 100 is best. A higher score indicates a better health state.
Time Frame: Baseline, Week 12
Population: Intent-to-treat, which consists of all patients who were randomized (started study) and received a baseline injection.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A 900kD | Placebo
Number analyzed (Participants) | 139 | 134
Scores on a Scale
  Baseline | 48.81 (9.70) | 46.40 (10.28)
  Week 12 | 51.16 (9.10) | 49.86 (9.82)

8. Secondary Outcome: Activities of Daily Living Quality of Life (QOL) Score at Week 24
Description: Activities of daily living QOL score at week 24 (or 10 weeks post second injection) as measured by SF-12 Physical Component (PCS-12). The SF-12 consists of 12 questions on various health questions. The PCS-12 is a sub-score calculated from the SF-12 total score based on the physical health questions where 0 is worse and 100 is best. A higher score indicates a better health state.
Time Frame: Baseline, Week 24
Population: Intent-to-treat, which consists of all patients who were randomized (started study) and received a baseline injection.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A 900kD | Placebo
Number analyzed (Participants) | 139 | 134
Scores on a Scale
  Baseline | 48.81 (9.70) | 46.40 (10.28)
  Week 24 | 52.34 (10.03) | 49.22 (10.36)

9. Secondary Outcome: Activities of Daily Living Quality of Life (QOL) Score at Week 52
Description: Activities of daily living QOL score at week 52 as measured by SF-12 Physical Component (PCS-12). The SF-12 consists of 12 questions on various health questions. The PCS-12 is a sub-score calculated from the SF-12 total score based on the physical health questions where 0 is worse and 100 is best. A higher score indicates a better health state.
Time Frame: Baseline, Week 52
Population: Intent-to-treat, which consists of all patients who were randomized (started study) and received a baseline injection.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A 900kD | Placebo
Number analyzed (Participants) | 139 | 134
Scores on a Scale
  Baseline | 48.81 (9.70) | 46.40 (10.28)
  Week 52 | 51.90 (9.44) | 50.34 (10.03)

10. Secondary Outcome: Direct Costs for Canada
Description: Direct healthcare costs associated with spasticity in cases where the primary reason for the use of the identified health care resource was the treatment of spasticity, or any related complications. Direct healthcare costs are presented in the local currency for Canada.
Time Frame: 52 Weeks
Population: Intent-to-treat, which consists of all patients in Canada who were randomized (started study) and received a baseline injection.
Measure: Mean (Standard Deviation); unit: Canadian dollar (CAD)
Arm/Group | Botulinum Toxin Type A 900kD | Placebo
Number analyzed (Participants) | 12 | 10
Canadian dollar (CAD) | 18643 (15022.4) | 13279 (10827.9)

11. Secondary Outcome: Direct Costs for Germany
Description: Direct healthcare costs associated with spasticity in cases where the primary reason for the use of the identified health care resource was the treatment of spasticity, or any related complications. Direct healthcare costs are presented in the local currency for Germany.
Time Frame: 52 Weeks
Population: Intent-to-treat, which consists of all patients in Germany who were randomized (started study) and received a baseline injection.
Measure: Mean (Standard Deviation); unit: Euro (EUR)
Arm/Group | Botulinum Toxin Type A 900kD | Placebo
Number analyzed (Participants) | 34 | 34
Euro (EUR) | 10181 (8110.1) | 10346 (7468.6)

12. Secondary Outcome: Direct Costs for Sweden
Description: Direct healthcare costs associated with spasticity in cases where the primary reason for the use of the identified health care resource was the treatment of spasticity, or any related complications. Direct healthcare costs are presented in the local currency for Sweden.
Time Frame: 52 Weeks
Population: Intent-to-treat, which consists of all patients in Sweden who were randomized (started study) and received a baseline injection.
Measure: Mean (Standard Deviation); unit: Swedish Krona (SEK)
Arm/Group | Botulinum Toxin Type A 900kD | Placebo
Number analyzed (Participants) | 48 | 44
Swedish Krona (SEK) | 93916 (75122.3) | 79580 (74951.3)

13. Secondary Outcome: Direct Costs for the United Kingdom
Description: Direct healthcare costs associated with spasticity in cases where the primary reason for the use of the identified health care resource was the treatment of spasticity, or any related complications. Direct healthcare costs are presented in the local currency for the United Kingdom.
Time Frame: 52 Weeks
Population: Intent-to-treat, which consists of all patients in the United Kingdom who were randomized (started study) and received a baseline injection.
Measure: Mean (Standard Deviation); unit: British Pound (GBP)
Arm/Group | Botulinum Toxin Type A 900kD | Placebo
Number analyzed (Participants) | 45 | 46
British Pound (GBP) | 4671 (6116.6) | 3977 (4039.2)

ADVERSE EVENTS:
Description: The Safety Population included all patients who were randomized and received at least 1 injection
Arm/Group | Botulinum Toxin Type A 900kD | Placebo
Serious Adverse Events (participants affected / at risk) | 47/139 | 45/134
Other Adverse Events (participants affected / at risk) | 60/139 | 45/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A 900kD (N=139) | Placebo (N=134)
Anaemia Megaloblastic (Blood and lymphatic system disorders) | 1 | 0
Angina Pectoris (Cardiac disorders) | 0 | 2
Atrial Fibrillation (Cardiac disorders) | 1 | 1
Cardiac Failure (Cardiac disorders) | 1 | 2
Left Ventricular Failure (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 2
Myocardial Ischaemia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Gastric Ulcer (Gastrointestinal disorders) | 1 | 0
Adverse Drug Reaction (General disorders) | 0 | 1
Non-cardiac Chest Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1
Escherichia Infection (Infections and infestations) | 1 | 0
Labyrinthitis (Infections and infestations) | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 2 | 4
Sepsis (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 2 | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 2 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 1 | 1
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 | 1
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 1
Polymyalgia Rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral Infarction (Nervous system disorders) | 1 | 2
Cerebrovascular Accident (Nervous system disorders) | 1 | 1
Cognitive Disorder (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 3 | 1
Depressed Level of Consciousness (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 2
Epilepsy (Nervous system disorders) | 2 | 4
Hemiparesis (Nervous system disorders) | 1 | 0
Lacunar Infarction (Nervous system disorders) | 1 | 0
Muscle Spasticity (Nervous system disorders) | 1 | 0
Partial Seizures (Nervous system disorders) | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 1
Urinary Retention (Renal and urinary disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Swelling Face (Skin and subcutaneous tissue disorders) | 1 | 0
Circulatory Collapse (Vascular disorders) | 0 | 2
Haematoma (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Temporal Arteritis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A 900kD (N=139) | Placebo (N=134)
Nasopharyngitis (Infections and infestations) | 13 | 11
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 8
Urinary Tract Infection (Infections and infestations) | 12 | 7
Fall (Injury, poisoning and procedural complications) | 18 | 15
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 7 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 7 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less